CLINICAL TRIAL: NCT01948869
Title: An Investigator-blinded, Randomized, Monocentre, 3-arm, Pilot Trial to Compare the Efficacy and Safety of Two Topical Medical Devices in Patients With Mild to Moderate Atopic Dermatitis in an Intra-individual Comparison With Untreated Skin
Brief Title: Efficacy/Safety Study to Explore a New Revised Topical Formulation in Atopic Dermatitis
Acronym: Phoenix II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16960; 2013-002569-20 (EudraCT Number)
Record Dates: First submitted 2013-09-19; First posted 2013-09-24 (Estimated); Last update posted 2014-08-07 (Estimated); Status verified 2014-08

CONDITIONS: Dermatitis, Atopic
Keywords: Phoenix; Mild atopic dermatitis; efficacy; safety
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Phoenix II (Experimental): Application over 29 days twice daily
  Interventions: Device: Phoenix II (BAY81-2996)
- Phoenix I (Active Comparator): Application over 29 days twice daily
  Interventions: Device: Phoenix I (BAY81-2996)
- Untreated skin (No Intervention): Untreated skin areas of subjects will be observed over 29 days

INTERVENTIONS:
Device: Phoenix II (BAY81-2996)
  Arms: Phoenix II
Device: Phoenix I (BAY81-2996)
  Arms: Phoenix I

SUMMARY:
The study shall explore whether treatment of atopic dermatitis is equally effective with respect to a marketed medical device and a new medical device.

ELIGIBILITY:
Inclusion Criteria:

* Male or female Caucasians aged between 18 and 60 years
* Patients with mild to moderate AD (Atopic Dermatitis) presenting a scoring AD (SCORAD) rating below 50
* Skin type I - IV according to Fitzpatrick
* Acute AD symptoms on each assessment areas (local SCORAD ≥ 3 and </= 12) at Baseline
* Acute symptom of pruritus at Baseline

Exclusion Criteria:

* Any other skin disease at the test area that would interfere the clinical assessment in the opinion of the investigator
* Moles, tattoos, strong pigmentation, or scars at the test area that would interfere the clinical assessment
* Regular intake of antiphlogistic drugs (for example, nonsteroidal anti-inflammatory drug [NSAIDs])
* Any condition or treatment which might influence the trial (e.g. any treatment with topical antibiotics, antifungals, or corticoids) within 14 days prior to screening as well as during the trial (exception: topical treatment of AD lesions other than the test areas (for example, face) with low potency steroids restricted to small areas)
* UV-therapy or the use of solarium within 30 days before screening as well as during the trial
* Any alternative treatment of AD (e.g. acupuncture, kinesiology, and homoeopathy) within 30 days before screening as well as during the trial

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2013-10; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Local scored atopic dermatitis (SCORAD) as clinical assessment by means of the intensity items of the SCORAD index | Up to 29 days

SECONDARY OUTCOMES:
Number of subjects with abnormal vital signs | Up to 10 weeks
  Vital signs consist of blood pressure, heart rate, and body temperature
Number of patients with adverse events as a measure of safety and tolerability | Up to 10 weeks
Erythema by means of chromametry | Up to 29 days
Transepidermal water loss (TEWL) as a measure for skin barrier function | Up to 29 days
Skin hydration by means of corneometry | Up to 29 days
Intensity of pruritus by means of visual analogue scale (VAS) | Up to 29 days

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Münster, North Rhine-Westphalia, Germany